CLINICAL TRIAL: NCT02766608
Title: A Randomized, Double-Blind, Parallel Group, Multi-Center Study to Assess the Efficacy and Safety of PT009 Compared to PT005, PT008, and Open-label Symbicort® Turbuhaler®, as an Active Control, on Lung Function Over a 24-Week Treatment Period in Subjects With Moderate to Very Severe COPD
Brief Title: Study to Assess Efficacy and Safety of PT009 Compared to PT005, PT008, and Symbicort® Turbuhaler® on Lung Function Over 24-Weeks in Subjects With Moderate to Very Severe COPD
Acronym: telos
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT009002
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disorder
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BFF MDI 320/9.6 μg (Experimental): Budesonide and Formoterol Fumarate Inhalation Aerosol 160/4.8 μg per actuation MDI/120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: BFF MDI 320/9.6 μg
- BFF MDI 160/9.6 μg (Experimental): Budesonide and Formoterol Fumarate Inhalation Aerosol-80/4.8 μg per actuation MDI/120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: BFF MDI 160/9.6 μg
- FF MDI 9.6 μg (Experimental): Formoterol Fumarate Inhalation Aerosol-4.8 μg per actuation MDI/ 120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: FF MDI 9.6 μg
- BD MDI 320 μg (Experimental): Budesonide inhalation Aerosol 160 μg per actuation MDI/120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: BD MDI 320 μg
- Symbicort® TBH 400/12 μg (Other): Symbicort Turbuhaler 400/12 μg Taken as 2 inhalations BID
  Interventions: Drug: Symbicort® TBH 400/12 μg BID

INTERVENTIONS:
Drug: BFF MDI 320/9.6 μg — Blinded Treatment
  Other Names: Budesonide and Formoterol Fumarate Inhalation Aerosol
  Arms: BFF MDI 320/9.6 μg
Drug: BFF MDI 160/9.6 μg — Blinded Treatment
  Other Names: Budesonide and Formoterol Fumarate Inhalation Aerosol
  Arms: BFF MDI 160/9.6 μg
Drug: FF MDI 9.6 μg — Blinded Treatment
  Other Names: Formoterol Fumarate Inhalation Aerosol
  Arms: FF MDI 9.6 μg
Drug: BD MDI 320 μg — Blinded Treatment
  Other Names: Budesonide Inhalation Aerosol
  Arms: BD MDI 320 μg
Drug: Symbicort® TBH 400/12 μg BID — Open Label
  Other Names: Symbicort® Turbuhaler
  Arms: Symbicort® TBH 400/12 μg

SUMMARY:
This is a Phase III randomized, double-blind, parallel group, multi-center, 24-week lung function study with BFF MDI (320/9.6 μg and 160/9.6 μg) compared to FF MDI 9.6 μg, BD MDI 320 μg, and open-label Symbicort® TBH (200/6 μg) administered BID.

DETAILED DESCRIPTION:
This is a Phase III randomized, double-blind, parallel group, multi-center, 24-week lung function study with BFF MDI (320/9.6 μg and 160/9.6 μg) compared to FF MDI 9.6 μg, BD MDI 320 μg, and open-label Symbicort® TBH (200/6 μg) administered BID. Subjects will undergo a 1- to 4-week Screening Period. Subjects who successfully complete the Screening Period will be to one of the following five treatment groups:BFF MDI 320/9.6 μg BID (N=660), BFF MDI 160/9.6 μg BID, FF MDI 9.6 μg BID, BD MDI 320 μg BID, Symbicort®, TBH 400/12 μg BID. Following randomization, subjects will enter the Treatment Period and undergo additional treatment visits over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Give their signed written informed consent to participate
2. Are at least 40 years of age and no older than 80 years
3. COPD patients who are symptomatic
4. Must be receiving one or more inhaled bronchodilators as maintenance therapy

Exclusion Criteria:

1. Current diagnosis of asthma,
2. COPD due to α1-Antitrypsin Deficiency
3. Known active tuberculosis, lung cancer, cystic fibrosis, significant bronchiectasis, Pulmonary resection or Lung Volume Reduction Surgery during the past 6 months
4. Long-term-oxygen therapy (≥ 12 hours a day).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2389 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (194):
- United States (73):
  - Research Site, Athens, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Gold River, California
  - Research Site, Palm Springs, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Boulder, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Hamden, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Panama City, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Blue Ridge, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Towson, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Jackson Heights, New York
  - Research Site, Larchmont, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Grove City, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Channelview, Texas
  - Research Site, Live Oak, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, South Burlington, Vermont
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Tacoma, Washington
- Canada (17):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Truro, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Mirabel, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Victoriaville, Quebec
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Québec
- Czechia (14):
  - Research Site, Boskovice
  - Research Site, Brandýs nad Labem
  - Research Site, Jindřichův Hradec
  - Research Site, Liberec
  - Research Site, Lovosice
  - Research Site, Nový Bor
  - Research Site, Ostrava-Hrabuvka
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
  - Research Site, Teplice
  - Research Site, Varnsdorf
  - Research Site, Žatec
- Germany (11):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Rodgau-Dudenhofen
  - Research Site, Schwerin
- Hungary (16):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Csorna
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Hatvan
  - Research Site, Komárom
  - Research Site, Makó
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Szolnok
- Poland (34):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Chełm
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Katowice
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Nowy Duninów
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Ostrów Wielkopolski
  - Research Site, Piekary Śląskie
  - Research Site, Piła
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Puławy
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Siedlce
  - Research Site, Sochaczew
  - Research Site, Suwałki
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Trzebnica
  - Research Site, Warsaw
  - Research Site, Wieluń
  - Research Site, Wołomin
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zamość
- Russia (23):
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Pytigorsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Ulyanovsk
  - Research Site, Vladimir
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Korea (6):
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- [Derived] Ferguson GT, Papi A, Anzueto A, Kerwin EM, Cappelletti C, Duncan EA, Nyberg J, Dorinsky P. Budesonide/formoterol MDI with co-suspension delivery technology in COPD: the TELOS study. Eur Respir J. 2018 Sep 16;52(3):1801334. doi: 10.1183/13993003.01334-2018. Print 2018 Sep. PMID 30220648
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4181&filename=PT009002_TELOS_PROTOCOL_REDACTED_07AUG2018_PDFA.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4181&filename=d7820c00001-12-1-09-Final_sap_PDFA.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4181&filename=PT009002_TELOS_PROTOCOL_REDACTED_PDFA.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4181&filename=PT009002_Final_sap_Redacted_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized subjects at 244 study centers in 7 countries, from June 2016 and November 2017. The study period was scheduled to take up to approximately 30 weeks for each individual subject from the time of screening through the follow-up period.
Pre-assignment Details: Subjects were randomized in a 3:3:3:1:1 ratio to BFF 320/9.6, BFF 160/9.6, FF 9.6, BD 320, and Symbicort.
Groups:
- BFF MDI 320/9.6 μg: Budesonide Formoterol Fumarate Metered Dose Inhalation 320/9.6 μg
- BFF MDI 160/9.6 μg: Budesonide Formoterol Fumarate Metered Dose Inhalation 160/9.6 μg
- FF MDI 9.6 μg: Formoterol Fumarate Metered Dose Inhalation 9.6 μg
- BD MDI 320 μg: Budesonide Metered Dose Inhalation 320 μg
- Symbicort TBH 400/12 μg: Symbicort Turbuhaler 400/12 μg
Period: Overall Study
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Started (mITT Population) | 655 | 637 | 644 | 206 | 219
Completed (Completed Treatment) | 576 | 567 | 554 | 169 | 190
Not Completed | 79 | 70 | 90 | 37 | 29
Not completed — Adverse Event | 27 | 22 | 17 | 13 | 12
Not completed — Withdrawal by Subject | 21 | 20 | 24 | 13 | 10
Not completed — Lack of Efficacy | 16 | 15 | 32 | 8 | 2
Not completed — Lost to Follow-up | 6 | 3 | 5 | 2 | 2
Not completed — Physician Decision | 3 | 2 | 3 | 1 | 2
Not completed — Protocol disc criteria | 3 | 3 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 4 | 0 | 1
Not completed — Administrative Reasons | 3 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Modified Intent-To-Treat (mITT) Population is a subset of the ITT Population, and is defined as all subjects with post-randomization data obtained prior to discontinuation from treatment. The Intent-To-Treat (ITT) Population is defined as all subjects who were randomized to treatment and received any amount of the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg | Total
Number analyzed (Participants) | 664 | 649 | 648 | 209 | 219 | 2389
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: mITT
  Years
    number analyzed (Participants) | 655 | 637 | 644 | 206 | 219 | 2361
    (all) | 64.2 (7.7) | 64.3 (7.6) | 64.1 (8.0) | 64.2 (7.4) | 65.3 (7.0) | 64.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: mITT
  Participants
    Values listed are mITT population: number analyzed (Participants) | 655 | 637 | 644 | 206 | 219 | 2361
    Values listed are mITT population: Female | 253 | 260 | 261 | 81 | 78 | 933
    Values listed are mITT population: Male | 402 | 377 | 383 | 125 | 141 | 1428
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT
  Participants
    Values listed are mITT population: number analyzed (Participants) | 655 | 637 | 644 | 206 | 219 | 2361
    Values listed are mITT population: Hispanic or Latino | 16 | 18 | 21 | 8 | 6 | 69
    Values listed are mITT population: Not Hispanic or Latino | 637 | 616 | 623 | 198 | 212 | 2286
    Values listed are mITT population: Unknown or Not Reported | 2 | 3 | 0 | 0 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT
  Participants
    Values listed are mITT population: number analyzed (Participants) | 655 | 637 | 644 | 206 | 219 | 2361
    Values listed are mITT population: American Indian or Alaska Native | 2 | 2 | 2 | 0 | 0 | 6
    Values listed are mITT population: Asian | 1 | 1 | 0 | 0 | 1 | 3
    Values listed are mITT population: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Values listed are mITT population: Black or African American | 19 | 15 | 20 | 9 | 8 | 71
    Values listed are mITT population: White | 633 | 619 | 622 | 197 | 210 | 2281
    Values listed are mITT population: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Values listed are mITT population: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 at Week 24 (BFF MDI Versus FF MDI)
Description: Change from baseline in morning pre-dose trough FEV1 (Forced expiratory volume in 1 second) at Week 24 (BFF MDI versus FF MDI)
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg
Number analyzed (Participants) | 571 | 564 | 550
Liter | 0.036 [0.019 to 0.053] | 0.017 [0.000 to 0.034] | -0.003 [-0.020 to 0.015]

2. Primary Outcome: Change From Baseline in FEV1 AUC0-4 (BFF MDI vs BD MDI)
Description: Changes from baseline in FEV1 AUC0-4 were normalized by taking the area under the curve value and dividing by the length of time under consideration (usually 4 hours). This normalization represents a weighted average of the change from baseline in FEV1 over the 4-hour period.
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Groups:
- FF MDI 9.6 ug: Formoterol Fumarate Metered Dose Inhalation 9.6 μg
- BD MDI 320 ug: Budesonide Metered Dose Inhalation 320 μg
- Symbicort TBH 400/12 ug: Symbicort Turbuhaler 400/12 ug
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 ug | BD MDI 320 ug | Symbicort TBH 400/12 ug
Number analyzed (Participants) | 571 | 565 | 549 | 168 | 189
Liter | 0.194 [0.177 to 0.212] | 0.179 [0.161 to 0.197] | 0.161 [0.143 to 0.179] | 0.022 [-0.011 to 0.054] | 0.187 [0.157 to 0.218]

3. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation (BFF MDI vs FF MDI).
Description: Time to first moderate or severe COPD (Chronic Obstructive Pulmonary Disease) exacerbation (BFF MDI vs FF MDI).
Time Frame: over 24 Weeks (timepoints of 4, 12 & 20 weeks)
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 ug
Number analyzed (Participants) | 655 | 637 | 644 | 206 | 219
Percentage of Participants
  Percentage of Subjects to Exacerbate at 4 Weeks | 3.2 [2.1 to 4.9] | 3.3 [2.2 to 5.1] | 5.5 [4.0 to 7.6] | 7.0 [4.2 to 11.5] | 1.8 [0.7 to 4.8]
  Percentage of Subjects to Exacerbate at 12 Weeks | 9.8 [7.7 to 12.4] | 9.9 [7.8 to 12.5] | 15.0 [12.4 to 18.1] | 14.9 [10.6 to 20.7] | 8.6 [5.5 to 13.3]
  Percentage of Subjects to Exacerbate at 20 Weeks | 14.4 [11.9 to 17.4] | 18.5 [15.6 to 21.8] | 20.5 [17.5 to 23.9] | 17.7 [13.0 to 23.9] | 13.1 [9.2 to 18.6]

4. Secondary Outcome: Percentage of Subjects Achieving an MCID (Minimal Clinically Important Difference) of 4 Units or More in SGRQ at Week 24
Description: The SGRQ (St. George's Respiratory Questionnaire) is a disease-specific questionnaire, self-completed by participants, used to evaluate the effect of BFF MDI, FF MDI, BD MDI, & Symbicort TBH on health-related quality of life as compared to placebo in subjects with COPD. The scores range from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Change from Baseline at a particular visit was calculated as the SGRQ total score at that visit minus Baseline. Change from Baseline in total score of -4 units or lower is considered as clinically meaningful improvement in quality of life.
Time Frame: at Week 24
Population: mITT
Measure: Number; unit: Percentage of Subjects
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 649 | 635 | 640 | 204 | 217
Percentage of Subjects | 48.12 | 47.22 | 41.59 | 43.62 | 53.78

5. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 at Week 24 (BFF MDI vs BD MDI)
Description: Change from baseline in morning pre-dose trough FEV1(Forced Expiratory Volume in 1 second) at Week 24 (BFF MDI vs BD MDI)
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 571 | 564 | 550 | 168 | 189
Liter | 0.036 [0.019 to 0.053] | 0.017 [0.000 to 0.034] | -0.003 [-0.020 to 0.015] | -0.028 [-0.060 to 0.003] | 0.039 [0.009 to 0.069]

6. Secondary Outcome: Peak Change From Baseline in FEV1 at Week 24 (BFF MDI vs BD MDI)
Description: Peak change from baseline in FEV1 (Forced Expiratory Volume in 1 second) at Week 24 (BFF MDI vs BD MDI)
Time Frame: at Week 24
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 571 | 565 | 549 | 168 | 189
Liter | 0.272 [0.254 to 0.291] | 0.258 [0.239 to 0.276] | 0.243 [0.224 to 0.261] | 0.116 [0.082 to 0.150] | 0.267 [0.253 to 0.299]

7. Secondary Outcome: Change From Baseline in Average Daily Rescue Ventolin HFA Use Over 24 Weeks (BFF MDI vs BD MDI)
Description: Change from baseline in average daily rescue Ventolin HFA use over 24 weeks (BFF MDI vs BD MDI)
Time Frame: over 24 Weeks
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs per day
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 654 | 636 | 641 | 206 | 218
Puffs per day | -1.3 [-1.5 to -1.1] | -1.3 [-1.4 to -1.1] | -1.1 [-1.2 to -0.9] | -0.6 [-0.9 to -0.3] | -1.2 [-1.5 to -0.9]

8. Secondary Outcome: FEV1 on Day 1, 5 Minutes, Time to Onset of Action Determination
Description: Time to onset of action Day 1 was evaluated by calculating change from baseline in FEV1 at each post-dose timepoint (5min, 15min, 30min, 1hr, 2hr, and 4hr), then comparing each treatment to BD MDI 320 ug. The first timepoint a statistically significant difference from BD MDI 320 ug of ≥100mL was determined to be time of onset for that treatment.
Time Frame: Day 1 - 5 Minutes
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 535 | 536 | 534 | 171 | 173
Liter | 0.157 [0.148 to 0.166] | 0.151 [0.142 to 0.161] | 0.160 [0.150 to 0.169] | 0.025 [0.009 to 0.041] | 0.131 [0.115 to 0.148]

9. Secondary Outcome: FEV1 on Day 1, 15 Minutes, Time to Onset of Action Determination
Description: as for outcome 8
Time Frame: Day 1 - 15 Minutes
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 624 | 615 | 612 | 203 | 211
Liter | 0.190 [0.180 to 0.200] | 0.186 [0.176 to 0.196] | 0.201 [0.191 to 0.211] | 0.040 [0.022 to 0.058] | 0.167 [0.149 to 0.184]

10. Secondary Outcome: FEV1 on Day 1, 30 Minutes, Time to Onset of Action Determination
Description: as for outcome 8
Time Frame: Day 1 - 30 Minutes
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 648 | 627 | 638 | 203 | 214
Liter | 0.207 [0.196 to 0.217] | 0.207 [0.196 to 0.218] | 0.215 [0.205 to 0.226] | 0.047 [0.028 to 0.066] | 0.190 [0.172 to 0.209]

11. Secondary Outcome: FEV1 on Day 1, 1 Hour, Time to Onset of Action Determination
Description: as for outcome 8
Time Frame: Day 1 - 1 Hour
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 649 | 628 | 640 | 204 | 215
Liter | 0.225 [0.213 to 0.236] | 0.221 [0.210 to 0.233] | 0.236 [0.225 to 0.248] | 0.053 [0.033 to 0.073] | 0.211 [0.191 to 0.231]

12. Secondary Outcome: FEV1 on Day 1, 2 Hours, Time to Onset of Action Determination
Description: as for outcome 8
Time Frame: Day 1 - 2 Hours
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 649 | 629 | 636 | 205 | 217
Liter | 0.253 [0.241 to 0.265] | 0.234 [0.222 to 0.247] | 0.244 [0.231 to 0.256] | 0.063 [0.042 to 0.085] | 0.221 [0.200 to 0.243]

13. Secondary Outcome: FEV1 on Day 1, 4 Hours, Time to Onset of Action Determination
Description: as for outcome 8
Time Frame: Day 1 - 4 Hours
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
Number analyzed (Participants) | 651 | 630 | 634 | 201 | 217
Liter | 0.230 [0.216 to 0.243] | 0.215 [0.202 to 0.229] | 0.212 [0.199 to 0.226] | 0.073 [0.049 to 0.097] | 0.209 [0.186 to 0.232]

14. Other Pre Specified Outcome: Substudy: 12-hour PFT Endpoint FEV1 AUC0-12
Description: Substudy: 12-hour PFT (Pulmonary Function Test) endpoint FEV1 (Forced Expiratory Volume) AUC0-12 (Area under the Curve 0-12). Changes from baseline in FEV1 AUC0-12 were normalized by taking the area under the curve value and dividing by the length of time under consideration. This normalization represents a weighted average of the change from baseline in FEV1 over the 12-hour period.
Time Frame: at Week 12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg
Number analyzed (Participants) | 160 | 167 | 189 | 47
Liter | 0.135 [0.107 to 0.163] | 0.124 [0.097 to 0.152] | 0.117 [0.089 to 0.145] | 0.024 [-0.028 to 0.075]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent throughout the treatment period and up to 14 days following the last dose of study drug
Description: Serious Adverse Events were collected from the time the subject signed informed consent throughout the treatment period and up to approximately 30 weeks, which includes screening and follow up (14 days after last dose of study drug).
Arm/Group | BFF MDI 320/9.6 μg | BFF MDI 160/9.6 μg | FF MDI 9.6 μg | BD MDI 320 μg | Symbicort TBH 400/12 μg
All-Cause Mortality (participants affected / at risk) | 3/655 | 2/637 | 2/644 | 0/206 | 2/219
Serious Adverse Events (participants affected / at risk) | 42/655 | 45/637 | 72/644 | 15/206 | 20/219
Other Adverse Events (participants affected / at risk) | 240/655 | 201/637 | 219/644 | 75/206 | 57/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 320/9.6 μg (N=655) | BFF MDI 160/9.6 μg (N=637) | FF MDI 9.6 μg (N=644) | BD MDI 320 μg (N=206) | Symbicort TBH 400/12 μg (N=219)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 10 (10) | 29 (35) | 2 (2) | 6 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5) | 6 (7) | 0 (0) | 3 (3)
Abdominal hernia gangrenous (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device battery issue (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 320/9.6 μg (N=655) | BFF MDI 160/9.6 μg (N=637) | FF MDI 9.6 μg (N=644) | BD MDI 320 μg (N=206) | Symbicort TBH 400/12 μg (N=219)
Nasopharyngitis (Infections and infestations) | 40 (46) | 40 (44) | 43 (46) | 17 (18) | 14 (18)
Upper respiratory tract infection (Infections and infestations) | 25 (27) | 21 (24) | 20 (20) | 5 (7) | 3 (3)
Chronic obstructive pulmonary disease (Infections and infestations) | 16 (17) | 10 (10) | 30 (36) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 14 (14) | 22 (22) | 15 (15) | 5 (5) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 13 (14) | 18 (19) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 19 (27) | 8 (10) | 15 (15) | 3 (4) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 15 (15) | 15 (15) | 7 (7) | 0 (0)
Oral candidiasis (Infections and infestations) | 17 (18) | 14 (15) | 5 (6) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (11) | 9 (9) | 7 (7) | 3 (3)
Bronchitis (Infections and infestations) | 16 (17) | 7 (8) | 10 (10) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 10 (12) | 9 (10) | 12 (13) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 9 (9) | 9 (9) | 5 (6) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 13 (13) | 3 (3) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (15) | 6 (6) | 6 (7) | 0 (0) | 8 (8)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2) | 4 (4) | 5 (5) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 5 (5) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT02766608/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02766608/SAP_001.pdf